CLINICAL TRIAL: NCT06274450
Title: A Clinical Study on the Improvement of Skin and Living Conditions After Drinking Rosa Roxburghii and Pomegranate Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botanee Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C2202112
Record Dates: First submitted 2023-12-20; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Skin Laxity
Keywords: Skin conditions
MeSH Terms: conditions — Cutis Laxa; Skin Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drinks with active ingredients Rosa Roxburghii and Pomegranate (Experimental): Take drinks with active ingredients such as Rosa Roxburghii and Pomegranate. Drink every morning on an empty stomach, 20ml/2 sachets/day.
  Interventions: Combination Product: skin care product; Other: Drinks with active ingredients Rosa Roxburghii and Pomegranate
- Blank Group (Other): Not taking drinks
  Interventions: Combination Product: skin care product

INTERVENTIONS:
Combination Product: skin care product — Subjects are uniformly using skin care products provided by the sponsor during the test. Skin care product include: WINONA sensitiveness relieving moisturizing cleansing foam, WINONA sensitiveness relieving moisturizing lotion, WINONA anti-sensitive tolerance-extreme moisturizing cream
Other: Drinks with active ingredients Rosa Roxburghii and Pomegranate — Take drinks with active ingredients such as Rosa Roxburghii and Pomegranate. Drink every morning on an empty stomach, 20ml/2 sachets/day.
  Arms: Drinks with active ingredients Rosa Roxburghii and Pomegranate

SUMMARY:
The main objective of the study is to observe changes in the subjects' skin condition and life status after 8 weeks of drinking rosa roxburghii and pomegranate drinks.

This is a single-center, randomized, single-blind, controlled, 8-week (56-day) clinical study conducted in Chinese healthy women aged 25-45 years old who were offered a rosa roxburghii and pomegranate drink.

DETAILED DESCRIPTION:
The study population is 70 healthy Chinese women aged 25-45 years who report current problems with dryness, roughness, dullness, and lack of elasticity on their face. The subjects will be randomly divided into an experimental group and a control product group of 35 subjects each.

Subjects will be formally enrolled after site assessment and subsequent site visits and test product administration. During the test cycle, subjects in the test group will take Prickly Pear Pomegranate Drink with active ingredients for 8 weeks, while the control product group will not take any test product. In order to avoid the influence of different skincare products on the results, all subjects will be asked to use a basic skincare product with moisturising ingredients only, provided by the sponsor, for the duration of the test. The efficacy of the test products will be verified by comparing the changes in skin condition and lifestyle of the subjects in the experimental group before taking the test products and 4 weeks and 8 weeks after taking the test products, as well as by comparing the differences in skin condition and lifestyle between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. 25-45 years old, Chinese female;
2. The subject's self-reported facial problems such as dryness, roughness, dullness, and lack of elasticity;
3. The subject's BMI is between 18~24kg/m2;
4. After the doctor's clinical evaluation, there is at least one obvious pigmentation spot with an ITA° difference of more than 10° on the face and the surrounding adjacent skin, and the diameter is not less than 3mm (it cannot be freckles, pigmented nevi, etc. that are difficult to improve clinically using topical preparations);
5. Corneometer base measurement of facial skin moisture at 15~45 (Corneometer Unit, C.U.) Between;
6. Be in good health and free of any other chronic diseases other than skin problems or diseases being treated;
7. Voluntarily participate in the test and sign the informed consent form;
8. Willing to comply with all evaluation requirements;

Exclusion Criteria:

1. Those who have used products, health foods or drugs with antioxidant and anti-aging effects in the past 2 months;
2. Those who have used any products, health foods or drugs (such as hydroquinone preparations) that affect skin color in the past 2 months;
3. Those who have used tretinoin preparations or undergone medical aesthetic treatments such as chemical peels, lasers, and pulsed light at the test site in the past 3 months;
4. Those who are inevitably exposed to long-term sunlight;
5. Intending to become pregnant, or being pregnant or breastfeeding;
6. Have a history of alcoholism;
7. Have a history of allergies;
8. Participated in any clinical trial evaluation within 1 month;
9. Those who have applied any anti-inflammatory drugs to the test site within the past two months;
10. Those who have suffered from skin diseases (such as psoriasis, eczema, psoriasis, skin cancer, etc.);
11. patients with insulin-dependent diabetes;
12. Patients with asthma or other chronic respiratory diseases who are being treated;
13. Have taken/injected anti-allergic drugs in the past 1 month;
14. Patients who have received anti-cancer chemotherapy or immunotherapy patients within the past 6 months;
15. Have a serious internal medicine disease, have any other health problems or chronic diseases;
16. Coated with retinoids, A hydroxy acids, salicylic acids, hydroquinone within the past 3 months, or prescription drugs (antibiotics, retinoids, A hydroxy acids and steroids) in use within the past 6 months, oral contraceptives (if you have been taking the same contraceptive pills for the past 6 months, you can continue to take them);
17. Experts or professionals believe that there are other iatrogenic causes that affect the results of the review.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Changes in the skin hydration | Week0（Baseline）、Week4、Week8
  Obtain change of skin hydration by Corneometer.
Changes in the skin glossiness | Week0（Baseline）、Week4、Week8
  Obtain change of skin glossiness by Glossymeter.
Changes in the skin firmness | Week0（Baseline）、Week4、Week8
  Obtain change of skin firmness by cutometer.
Changes in the skin elasticity | Week0（Baseline）、Week4、Week8
  Obtain change of skin elasticity by cutometer.
Changes in the individual type angle | Week0（Baseline）、Week4、Week8
  Obtain change of Individual type angle by Colorimeter.
Changes in the melanin content | Week0（Baseline）、Week4、Week8
  Obtain change of melanin content by Mexameter MX18.
Changes in the proportion of crow's feet area | Week0（Baseline）、Week4、Week8
  Calculate the proportion of crow's feet area by Visia CR images.
Changes in the proportion of fine lines under the eye | Week0（Baseline）、Week4、Week8
  Calculate the proportion of fine lines under the eye by Visia CR images.
Changes in the CIE RGB of skin tone | Week0（Baseline）、Week4、Week8
  Dermatologist use PANTONE SkinTone (Pantone color card) skin color guide to evaluate skin tone grade of subjects. Find the CIE RGB corresponding to the skin tone grade in Pantone ColorManager software and convert it into a color value using the formula for data analysis: CIE RGB = R+G*256+B*256*256.
  Calculate the change of CIE RGB of skin tone.
Changes in the grade of Pigmentation | Week0（Baseline）、Week4、Week8
  Obtain change of degree of Pigmentation severity by Dermatologist evaluation according to Skin Aging ATLAS of Asian Type.
Skin condition Assessment after 4-week application | Week4
  Obtain data on agreement with skin condition improvement by skin condition self-assessment questionnaire. The questionnaire is a 9-point scale, with 1 indicating strong disagreement and 9 indicating strong agreement.
Skin condition Assessment after 8-week application | Week8
  Obtain data on agreement with skin condition improvement by skin condition self-assessment questionnaire. The questionnaire is a 9-point scale, with 1 indicating strong disagreement and 9 indicating strong agreement.

SECONDARY OUTCOMES:
Changes in the satisfaction with the quality of life | Week0（Baseline）、Week4、Week8
  Obtain change of satisfaction with the quality of life accessed by WHOQOL-100 questionnaire. The questionnaire is a 5-point scale, with 1 indicating very dissatisfied and 5 indicating very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Zhan Wang, Master, Principal Investigator — Shenzhen Fubiyu Clinic
Locations (1):
- Shanghai China-norm Quality Technical Service Co ，Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is used to develop new products, no decision has been made on when to disclose